CLINICAL TRIAL: NCT01041443
Title: A Phase I Study of 5-Fluoro-2'-Deoxycytidine With Tetrahydrouridine (FdCyd + THU) in Myeloid Leukemia and MDS
Brief Title: 5-Fluoro-2'-Deoxycytidine and Tetrahydrouridine in Treating Patients With Acute Myeloid Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09045; NCI-2009-01661
Record Dates: First submitted 2009-12-29; First posted 2009-12-31 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Adult Acute Myeloid Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 5-fluoro-2'-deoxycytidine; Tetrahydrouridine; Reverse Transcriptase Polymerase Chain Reaction; DNA Methylation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive FdCyd IV over 3 hours and THU IV over 3 hours on days 1-10. Courses repeat every 21days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 5-fluoro-2-deoxycytidine; Drug: tetrahydrouridine; Other: laboratory biomarker analysis; Genetic: reverse transcriptase-polymerase chain reaction; Genetic: DNA methylation analysis

INTERVENTIONS:
Drug: 5-fluoro-2-deoxycytidine — Given IV
  Other Names: FdCyd
Drug: tetrahydrouridine — Given IV
  Other Names: THU
Other: laboratory biomarker analysis — Correlative studies
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR
Genetic: DNA methylation analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of 5-Fluoro-2'-deoxycytidine (FdCyd) when given together with tetrahydrouridine (THU) in treating patients with acute myeloid leukemia (AML) or myelodysplastic syndromes (MDS). FdCyd may inhibit cancer cell growth by increasing the production in cells of compounds that suppress growth or by otherwise killing cells. Although FdCyd is stable as a drug solution, it is rapidly inactivated by an enzyme present in people. THU is included in the treatment to inhibit the enzyme, prolonging the time FdCyd remains in the body

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of FdCyd administered with a fixed dose of THU in patients with acute myelogenous leukemia (AML) and myelodysplastic syndrome (MDS), once daily on days 1-10 of a 21-day treatment cycle. II. To describe the toxicities of FdCyd/THU in patients with acute myelogenous leukemia (AML) and myelodysplastic syndrome (MDS). III. To document all clinical responses and hematologic improvement in patients treated with FdCyd/THU. IV. To obtain preliminary information regarding the effect of FdCyd/THU on deoxyribonucleic acid (DNA) methylation patterns in peripheral blood mononuclear cells and bone marrow aspirates, including malignant myeloid cells; the ratio of gamma- to beta-globin messenger ribonucleic acid (mRNA) in blood cells; and serum cytokines. OUTLINE: This is a dose-escalation study of FdCyd. Patients receive FdCyd intravenously (IV) over 3 hours and THU IV over 3 hours on days 1-10. Courses repeat every 21days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients must have the following diagnosis:

* Acute myeloid leukemia

  * Relapsed or refractory
  * Newly diagnosed in patients age 60 and above or of any age unable to receive standard induction regimen
* Patients with MDS with an International Prognostic Scoring System (IPSS) score >= 0.5

  * Newly diagnosed
  * Relapsed or refractory
* Any prior therapy must have been completed >= 2 weeks prior to enrollment and the participant must have recovered to eligibility levels from prior toxicity
* No limit to number of prior regimens
* Hydroxyurea is allowed prior to enrollment to keep white blood cell count (WBC) below 20 K
* Valproic acid not being used for seizure control should be stopped 72 hours before starting therapy
* Prior therapy with hypomethylating agent (decitabine or azacitidine) is allowed and must be completed >= 6 weeks prior to enrollment
* Relapsed patients are eligible post allogeneic or matched unrelated donor (MUD) transplant after 100 days; there should be no active acute graft versus host disease of any grade and patient should not be receiving immunosuppression for acute graft versus host disease; the patient must not have Chronic Graft versus Host disease (cGvHD) other than mild skin, oral, or ocular cGvHD not requiring systemic immunosuppression
* Relapsed patients are eligible post autologous transplant after 100 days post transplant, with recovery of their counts absolute neutrophil count (ANC) > 1000 and platelets greater than 75K at some point post transplant
* Karnofsky performance status >= 60%
* Total bilirubin < 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine < 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min for patients with creatinine levels above 1.5 x institutional upper limit of normal
* Pregnant women will be excluded from this trial; nursing women are also excluded; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation, and for 3 months after completion of study; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients should not be receiving any other investigational agents

Exclusion Criteria:

* Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to: active or uncontrolled infection, immune deficiencies or confirmed diagnosis of human immunodeficiency virus (HIV) infection, active Hepatitis B, active Hepatitis C, or uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with additional (other than AML/MDS) currently active primary malignancy other than curatively treated carcinoma in situ (CIS) of the cervix, or basal or squamous cell carcinoma of the skin; patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy and disease free from prior malignancies for > 2 years
* Patients with active central nervous system (CNS) disease; these patients are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Active infections, including opportunistic following allo, MUD, or auto transplant (including but not limited to cytomegalovirus [CMV], fungal infection etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
MTD and dose-limiting toxicity (DLT) of the new 10-day schedule of FdCyd/THU | 10 days
  Toxicities will be summarized by Common Terminology Criteria for Adverse Events (CTCAE) grade and attribution using the version current at the initiation of the protocol.

SECONDARY OUTCOMES:
Toxicities of the FdCyd/THU treatment | 3 years
Time to progression | 3 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chen, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States